CLINICAL TRIAL: NCT06607653
Title: The Efficacy of Olfactory Training Intervention on Olfactory and Other Non-motor Symptoms in PD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, WANG KAI, Head, Dept of Neurology & Medical Psychology, Director, Cognitive Neuropsychology Lab, PRC, Anhui Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AHMU-PD-OT
Record Dates: First submitted 2024-09-19; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease; Olfactory Disorder; Olfactory Training
Keywords: Parkinson Disease; Olfactory Disorder; Olfactory training
MeSH Terms: conditions — Parkinson Disease | interventions — Olfactory Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT grroup (Experimental): Olfactory training used repeated stimulation of different olfactory substances at high concentrations, combined with odor association and odor identification training, twice in the morning and evening, each time for 5 minutes, for 15 weeks.
  Interventions: Device: Olfactory training
- No intervention group (No Intervention): There were only pre-test and post-test without any intervention

INTERVENTIONS:
Device: Olfactory training — Olfactory training used repeated stimulation of different olfactory substances at high concentrations, combined with odor association and odor identification training, twice in the morning and evening, each time for 5 minutes, for 15 weeks.
  Arms: OT grroup

SUMMARY:
To explore the efficacy of olfactory training on olfactory and other non-motor symptoms in PD.

ELIGIBILITY:
Inclusion Criteria:

1. PD was diagnosed according to the criteria of Movement Disorders and Parkinson Disease Group of Chinese Society of Neurology of Chinese Medical Association.
2. Olfactory score was 1 standard deviation lower than the corresponding age norm;
3. no medication plan in the past four weeks or no change in medication plan in the past four weeks, which can be maintained until the end of the experiment; 4.40-75 years old, with normal vision, hearing and language understanding and expression ability;

5.Good cooperation of patients

Exclusion Criteria:

1. Parkinson's syndrome and Parkinson's plus syndrome caused by cerebrovascular disease, encephalitis, trauma, drugs, etc.;
2. Neuropsychiatric diseases that may affect the sense of smell, such as depression, anxiety, schizophrenia, etc.;
3. History of nasal disease or surgery, such as rhinitis, sinusitis, nasal septum deviation, etc. Upper respiratory tract infection in the past 3 weeks;
4. Long-term smoking and occupations that inhale chemical irritants for a long time.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-25 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Olfactory Function Test | baseline;15 weeks
  The olfactory test developed by the Institute of Psychology, Chinese Academy of Sciences was used to evaluate the olfactory ability, including threshold, discrimination, and recognition.

SECONDARY OUTCOMES:
MoCA | baseline;15 weeks
Pittsburgh sleep quality index | baseline;15 week
HAMA | baseline;15week
HAMD | baseline;15 week

CONTACTS AND LOCATIONS:
Locations (1):
- Cognitive Neuropsychology Lab Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No